CLINICAL TRIAL: NCT03392129
Title: Ai Chi Method for Children With Asthma: A Single-blinded Randomized Controlled Trial
Brief Title: Ai Chi Method for Children With Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Karla Morganna Pereira Pinto de Mendonça, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67253617.4.0000.5537
Record Dates: First submitted 2017-12-28; First posted 2018-01-05 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Asthma; Child; Respiratory Disease; Hydrotherapy; Respiratory Tract Diseases; Respiratory Hypersensitivity; Respiration Disorders
Keywords: Asthma; Child; respiratory exercises; Hydrotherapy; Physical Therapy Specialty; Sleep; Quality of life; Anxiety; Spirometry; Clinical trial
MeSH Terms: conditions — Asthma; Respiration Disorders; Respiratory Tract Diseases; Respiratory Hypersensitivity; Anxiety Disorders | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ai Chi (Experimental): Children in the intervention group will perform 12 sessions (twice a week, 40 minutes each session) of treatment with the Ai Chi Method and educational interventions in relation to asthma.
  Interventions: Other: Ai Chi
- Asthma education (Active Comparator): Children assigned to the control group will receive, along with their parents, educational interventions in relation to asthma.
  Interventions: Other: Asthma education

INTERVENTIONS:
Other: Ai Chi — Children in the intervention group will perform 12 sessions (twice a week 40 minutes each session) of treatment with the Ai Chi Method, and educational intervention in relation to asthma.
  Arms: Ai Chi
Other: Asthma education — Children assigned to the control group will receive, along with their parents, educational interventions in relation to asthma.
  Arms: Asthma education

SUMMARY:
This study has the aim to assess the effectiveness of the Ai Chi method as an adjunct therapy in the treatment of children with asthma.

DETAILED DESCRIPTION:
Children from 7 to 12 years old with asthma diagnosis will be included. Children assigned to the control group will receive, along with their parents, educational interventions in relation to asthma, based on guidelines of Global Strategy for Asthma Management and Prevention Revised 2017.Children in the intervention group will perform 12 sessions (twice a week) of treatment with the Ai Chi Method and educational interventions similiar to the control group. The investigators will assess pulmonary function (spirometry), asthma control by the Childhood Asthma Control Test (c-ACT Questionnaire), quality of life by the PAQLQ (Paediatric Asthma Quality of Life Questionnaire), anxiety symptoms by the SCAS (Spence Children's Anxiety Scale) and Disturbed Sleep by the Sleep Disorders Scale in Children. In addition, information will be collected on the numbers of hospitalizations, occurence of absence in school due to exacerbation of the disease, asthma symptoms and Beta2-agonists usage.

ELIGIBILITY:
Inclusion Criteria:

* Children from 7 up to 12 years old with asthma diagnose;
* Regular inhaled corticosteroids with no change in dose in the preceding 4 weeks;
* Children cannot present: other respiratory disease (such as cystic fibrosis, bronchiectasis, tuberculosis), obesity, retinal detachment, hypertensive crisis, congenital heart defect, pulmonary edema, history of lobectomy or lung segmentectomy, respiratory infections 15 days prior to the evaluations.

Exclusion Criteria:

* Children that are not able to perform some of the necessary procedures;
* Give up participating in the research and present acute symptoms of respiratory tract during the assessments.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-07-20 (Estimated); Study Completion 2020-07-20 (Estimated)

PRIMARY OUTCOMES:
Change in Lung function (spirometry). | Baseline, six weeks later (endpoint) and one month since the initial of intervention (follow-up)
  Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), FEV1/FVC ratio, forced expiratory flow between 25-75% of the pulmonary volume (FEF25-75).

SECONDARY OUTCOMES:
Change in asthma control. | Baseline, six weeks later (endpoint) and one month since the initial of intervention (follow-up)
  Asthma control will be assessed by the Childhood Asthma Control Test - c-ACT Questionnaire Mean c-ACT score. Do higher values of 19 points represent a better outcome .
Change in Quality of life | Baseline, six weeks later (endpoint) and one month since the initial of intervention (follow-up)
  Quality of life of childhood asthma as assessed by the Standardized Pediatric Asthma Quality of Life Questionnaire (PAQLQ). 7 point rating scale Do higher values represent a better outcome.
Change in Anxiety symptoms. | Baseline, six weeks later (endpoint) and one month since the initial of intervention (follow-up)
  Change in Spence Children's Anxiety Scale following intervention. Self-reported (child and parent version) child anxiety symptoms, 38 items questionnaire, rated at a 4-point scale. Do higher values represent a worse outcome.
Change in Disturbed Sleep. | Baseline, six weeks later (endpoint) and one month since the initial of intervention (follow-up)
  Disturbed Sleep will be assessed by the Sleep Disorders Scale in Children. 26 items questionnaire, rated at a 5-point scale. Do higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Karla Mendonça, PT, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte; Renata Tomaz, PT, PhD's Student, Principal Investigator — Universidade Federal do Rio Grande do Norte; Ada Jácome, PT, PhD's student, Principal Investigator — Universidade Federal do Rio Grande do Norte; Thayla Amorim, PT, Ms, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Universidade Federal do Rio Grande do Norte (UFRN), Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No